CLINICAL TRIAL: NCT01655407
Title: Evaluation of Autologous Engineered Skin Substitute (ESS-W) Compared to Meshed, Split-Thickness Autograft (AG) for Treatment of Deep Partial- and Full-Thickness Thermal Burn Wounds in Adult Patients
Brief Title: Safety and Efficacy Study of Autologous Engineered Skin Substitute to Treat Partial- and Full-Thickness Burn Wounds
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Amarantus BioScience Holdings, Inc. (Industry)
Collaborators: Amarex Clinical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Lonza-ESS01
Record Dates: First submitted 2012-07-20; First posted 2012-08-01 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Thermal Injury; Deep Partial-Thickness Burn; Full-Thickness Burn
Keywords: Split-thickness Autograft; Engraftment; Wound Closure; Engineered Skin Substitute; ESS-W; Cultured Skin Substitutes; Burn
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Experimental): All patients will receive both Autologous Engineered Skin Substitute (ESS-W) and Split-Thickness Autograft (AG).
  Interventions: Drug: Autologous Engineered Skin Substitute; Drug: Split-Thickness Autograft (AG)
- Control (Active Comparator): All patients will receive both Autologous Engineered Skin Substitute (ESS-W) and Split-Thickness Autograft (AG).
  Interventions: Drug: Autologous Engineered Skin Substitute; Drug: Split-Thickness Autograft (AG)

INTERVENTIONS:
Drug: Autologous Engineered Skin Substitute — The total burn wound area covered will range from 288 cm^2 to 5,600 cm^2 (based on availability of matched-pair burn sites of similar area and depth) and this total grafting area will be divided equally for treatment with ESS-W and AG.
  ESS-W will be applied to the appropriate recipient site, according to the randomization schedule, by the surgeon using two pairs of forceps. Sufficient ESS-W sheets will be used to cover the recipient site. The ESS-W grafts will be stapled in place.
  Other Names: ESS-W
Drug: Split-Thickness Autograft (AG) — The total burn wound area covered will range from 288 cm^2 to 5,600 cm^2 (based on availability of matched-pair burn sites of similar area and depth) and this total grafting area will be divided equally for treatment with ESS-W and AG.
  The AG regimen occurs in stages, beginning with excision of the burned skin, followed by temporary wound coverage (e.g. cadaveric skin allografts, porcine xenograft, synthetic or biologic dressings or medical devices) to achieve wound homeostasis, and completed by permanent wound closure using autologous skin.
  Other Names: Split-thickness skin grafts (STSGs)

SUMMARY:
The purpose of this research study is to test how well the investigational treatment, Engineered Skin Substitutes (ESS-W), works for covering and treating burn wounds.

The areas of the body that are treated with ESS-W will be compared to similar areas treated with the patient's own skin (split-thickness skin autograft (AG)). A skin autograft (AG) will be performed by taking healthy skin from one area of the body and placing it on the burned area.

DETAILED DESCRIPTION:
This study is designed to evaluate the safety and efficacy of autologous engineered skin substitute (ESS-W) compared to conventional split-thickness AG for the treatment of extensive, deep partial- and full-thickness thermal burns. A matched and randomized burn site format will be used to evaluate the successful graft take on excised deep partial- and full-thickness burns when grafted with either 1) unmeshed ESS-W or 2) meshed AG (the current standard treatment of split thickness AG).

This research study is divided into five study periods: (1) Screening Period of up to one week and (2) Pre-Grafting Period, which will last approximately 35-45 days, (3) Grafting Day(s), which are the day(s) on which grafts are applied (i.e., First Graft: Day 0 and the optional subsequent Grafting Day i.e., Second Graft: Day 0), (4) Post Grafting Observation Period, which begins with 28 days follow-up after each Grafting Day(s), and continues till Post-Operative Month (POM) 6 from the last Grafting Day, and (5) Anecdotal Observation Period

ELIGIBILITY:
Inclusion Criteria:

* Has deep partial or full-thickness thermal burns ≥50% of the TBSA and fulfills the total grafting area requirement ranging from 288 cm2 up to 5,600 cm2, divided between two (or more) recipient sites.
* Is expected to require multiple skin grafting procedures.
* Is ≥18 years and ≤40 years of age at the time of enrollment.
* Females of childbearing potential must have a negative pregnancy test prior to enrollment and agree to use appropriate birth control methods during the pre-grafting period and for three months following the last Grafting Day.
* Subject (or a legally authorized representative (LAR)) has provided written informed consent for study participation and procedures to be performed.

Exclusion Criteria:

* Has a current diagnosis of septic shock or Multiple Organ Dysfunction Syndrome, which in the opinion of the Investigator would put the potential subject at risk of serious morbidity or death by participating in the study.
* Has a current diagnosis of an invasive burn wound infection in unexcised burn wound.
* Is pregnant.
* Is a prisoner at the time of obtaining written informed consent.
* Has a documented history of allergy or sensitivity to any of the antimicrobials or reagents used in preparation and application of ESS-W including the irrigation solution used before and after grafting. These include aminoglycosides, polymyxin B, mupirocin, ciprofloxacin, amphotericin B, hydrocortisone, and insulin.
* Has a documented history of allergy or sensitivity to any of the animal products used in preparation of ESS-W. These products include bovine blood, bovine collagen, bovine collagenase, and porcine trypsin-versene.
* Has a documented history of allergy or sensitivity to glycosaminoglycan, the polymer component of ESS-W.
* Has a documented ongoing condition which could delay wound healing such as insulin-dependent diabetes mellitus, Cushing syndrome or disease, scurvy, chronic hypothyroidism, congenital or acquired immunosuppressive condition, chronic renal failure, or chronic hepatic dysfunction (Child-Pugh class B or C).
* Has a severe malnutrition or other concomitant illness which, in the opinion of the Investigator, has the potential to significantly delay wound healing.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-09; Primary Completion 2019-12 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of infections at grafting sites | Up to Month 6 after the last grafting day
  Assessments will be done on the following days/months:
  * Post operative Day 1 - Day 6, Day 7, Day 14 and Day 28 after each grafting day.
  * Post Operative Month 3 and Month 6 after the last grafting day.
Incidence of re-grafting | Up to Month 6 after the last grafting day
  Assessments will be done on the following days/months:
  * Post operative Day 7, Day 14 and Day 28 after each grafting day.
  * Post Operative Month 3 and Month 6 after the last grafting day.
Incidence of adverse events that are related to study treatment and associated with the grafting site | Up to Month 36 after the last grafting day
  Assessments will be done on the following days/months:
  * Post operative Day 1 - Day 6, Day 7, Day 14 and Day 28 after each grafting day.
  * Post Operative Month 3, Month 6, Month 12, Month 24 and Month 36 after the last grafting day
Incidence of all adverse events. | Up to Month 36 after the last grafting day
  Assessments will be done on the following days/months:
  * Post operative Day 1 - Day 6, Day 7, Day 14 and Day 28 after each grafting day.
  * Post Operative Month 3, Month 6, Month 12, Month 24 and Month 36 after the last grafting day
Percentage engraftment as determined by the Investigator through clinical assessment | Up to Month 3 after the last grafting day
  Assessments will be done on the following days/months:
  * Post operative Day 14 and Day 28 after each grafting day.
  * Post Operative Month 3 after the last grafting day
Percentage engraftment as determined by an independent observer through clinical assessment | Up to Month 3 after the last grafting day
  Assessments will be done on the following days/months:
  * Post operative Day 14 and Day 28 after each grafting day.
  * Post Operative Month 3 after the last grafting day
Confirmation of engraftment by histological assessment | Up to Month 6 after the last grafting day
  Assessments will be done on the following days/months:
  - Post Operative Month 3 and Month 6 after the last grafting day
Percentage of wound closure as determined by blinded computerized planimetric assessment | Up to Month 3 after the last grafting day
  Assessments will be done on the following days/months:
  * Post operative Day 14 and Day 28 after each grafting day.
  * Post Operative Month 3 after the last grafting day
Percentage area of re-grafting as determined by blinded computerized planimetric assessment | Up to Month 6 after the last grafting day
  Assessments will be done on the following days/months:
  * Post operative Day 7, Day 14 and Day 28 after each grafting day.
  * Post Operative Month 3 and Month 6 after the last grafting day.

SECONDARY OUTCOMES:
Scar outcome assessment using the modified Vancouver Scar Scale (mVSS). | Up to Month 36 after the last grafting day
  Assessments will be done on the following days/months:
  * Post operative Day 28 after each grafting day.
  * Post Operative Month 3, Month 6, Month 12, Month 24 and Month 36 after the last grafting day
Incidence and severity of post-burn pruritus utilizing a validated patient self-assessment instrument | Up to Month 36 after the last grafting day
  Assessments will be done on the following days/months:
  * Post operative Day 14 and Day 28 after each grafting day.
  * Post Operative Month 3, Month 6, Month 12, Month 24 and Month 36 after the last grafting day
Incidence of contracture release or revision surgeries | Up to Month 36 after the last grafting day
  Assessments will be done on the following days/months:
  - Post Operative Month 3, Month 6, Month 12, Month 24 and Month 36 after the last grafting day
Incidence of increased temperature sensitivity | Up to Month 36 after the last grafting day
  Assessments will be done on the following days/months:
  - Post Operative Month 3, Month 6, Month 12, Month 24 and Month 36 after the last grafting day
Incidence of paresthesias, pain, dulling of sensation assessed through patient self-reporting scale and by monofilament testing | Up to Month 36 after the last grafting day
  Assessments will be done on the following days/months:
  - Post Operative Month 3, Month 6, Month 12, Month 24 and Month 36 after the last grafting day

CONTACTS AND LOCATIONS:
Overall Officials: Michael Peck, MD, Study Director — The Arizona Burn Center
Locations (3):
- United States (3):
  - Arizona Burn Center, Pheonix, Arizona
  - US Army Institute of Surgical Research, Houston, Texas
  - Harborview Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided